CLINICAL TRIAL: NCT05527028
Title: Does Occupational Directed Services in Long-term Care Maintain a Resident's Self Performance in Activities of Daily Living: A Pilot Study
Brief Title: OT Directed Services in Long-term Care in Ontario
Acronym: OTLTC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Laurie Perrett, Director of Clinical Education, Occupational Therapy, McMaster University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 001
Record Dates: First submitted 2022-02-18; First posted 2022-09-02 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Aging

STUDY DESIGN:
Intervention Model Description: Pilot study for single site trial.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participant group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Both groups will receive the standard care provided at the long-term care home. The intervention group will receive the addition of directed occupational therapy intervention provided by student occupational therapists for up to 30 minutes, five days a week. At present, no decisive evidence exists that this intervention being tested will be superior to the standard of care.
  Interventions: Other: Occupational Therapy Services
- Intervention Group (Experimental): Both groups will receive the standard care provided at the long-term care home. The intervention group will receive the addition of directed occupational therapy intervention provided by student occupational therapists for up to 30 minutes, five days a week. At present, no decisive evidence exists that this intervention being tested will be superior to the standard of care.
  Interventions: Other: Occupational Therapy Services

INTERVENTIONS:
Other: Occupational Therapy Services — Investigators will complete an initial assessment based on a thorough chart review and observation of the participants activities of daily living during week one. The resident will receive approximately 30 minutes a day of direct student OT service delivery. Additional intervention may be delivered through an indirect, collaborative, or consultative service delivery model. Students will use a workload measurement tool to track the amount of time and types of intervention provided to these residents. The intervention will be delivered by two pairs of OT students under the direction of a registered OT. Student OTs will have access to Point Click Care and will document daily and will be required to document indirect and non-direct time for each resident.

SUMMARY:
In long-term care, staff provide help to residents with bathing, dressing, eating, walking, toileting, transferring, and moving in bed. Some residents can do more for themselves than others. This study will compare two groups of residents who require the same level of help from staff. Over eight weeks, one group will receive occupational therapy services provided by OT students and the other group will not. After the eight weeks, the level of help that each group of people requires will be looked at to see if there are any differences.

DETAILED DESCRIPTION:
A pilot study to determine if Occupational Therapy (OT) directed service in long-term care maintain a resident's self-performance in activities of daily living: Study protocol for a single-site trial

INTRODUCTION AND BACKGROUND

In Canada, a significant gap exists in providing resident-focused services to individuals in long-term care homes (LTCHs) to promote maintenance of function and participation in activities of daily living (McArthur et al., 2015; Ontario Society of Occupational Therapy, OSOT, 2020). People who live in LTCHs are frail, have some form of cognitive impairment, and live with at least one chronic health condition (McArthur et al., 2017; Ontario Long-Term Care Association, OLTCA, 2019, Shakeel et al., 2015). Upon admission to an LTCH, an alarming number of individuals experience a stark decline in function in activities of daily living (Crocker et al., 2013). Furthermore, the number of residents who require extensive assistance with activities of daily living (ADLs), such as grooming, getting dressed, and eating is also rising. For example, in 2018, 86% of long-term care residents in Ontario required extensive assistance with ADLs (OLTCA, 2019). However, this alarming trend may bring to question if this is an accurate representation of residents' true abilities or possibly the lack of resident-focused services that support a restorative care philosophy, in which allows individuals to maintain current abilities or decelerate functional decline after admission to LTC.

The lack of rehabilitation services in LTCHs is disturbing. Residents should have access to services that aim to prevent further rapid decline in function or participation in activities of daily living (ADLs). The LTCH Act in Ontario states that "Every resident has the right to receive care and assistance towards independence based on a restorative care philosophy to maximize independence to the greatest extent possible." (Long-Term Care Homes Acts, 2007, 2-3). Nationally, OT accounts for only 4.0% of the rehabilitation services presently provided within LTCHs. Ontario has the lowest percentage of LTCH residents' access to OT across Canada (Canadian Institute of Health Information, 2019). OT-directed services in LTCHs can address specific resident needs related to daily living activities by identifying and help to lessen risks residents are face with in LTCH, which often result in increased care demands for the LTCH team (OSOT, 2020). Evidently, long-term homes in Ontario are challenged to pilot alternative ways in which a restorative care approach can be modelled and delivered in LTC for residents to fulfill this mandate.

According to the 2021 Ontario budget announcement, the province pledged to increase the average direct care to four hours a day in long-term care and hire more than 27,000 new staff positions, including allied health professionals (Ontario Ministry of Finance, 2021). With this influx of new funding and additional human resources, the current delivery model of rehabilitation services in long-term care must be re-considered. Furthermore, a pilot to test an innovative model of OT-directed service delivery to facilitate a restorative care philosophy is necessary to maximize resident function and level of participation in daily activities.

A registered occupational therapist will direct student occupational therapists to assess and develop resident-focused interventions to be implemented and evaluated by the long-term care team. We seek to understand if OT-directed services delivered by student OTs will demonstrate maintenance of function in long-term care home residents.

We propose a two-phase study that will use a pilot design first to test the ability to identify eligible residents, implement the model, and assess outcomes (Pilot Study), which will inform the design of a more extensive outcomes study (Main Trial).

1.2 PILOT OBJECTIVES AND RESEARCH QUESTIONS

The objectives of the Pilot Study will be to determine if:

* Potential participants can be identified and are willing consent to the Pilot Study
* If the intervention can be implemented as intended
* Outcomes can be measured consistently

PRIMARY RESEARCH QUESTION: Will the provision of occupational therapy intervention, provided by student occupational therapists for 30 minutes a day for eight weeks, maintain resident performance in activities of daily living in long-term care as reported using the Modified Barthel Index?

SECONDARY RESEARCH QUESTION:

Does the provision of occupational therapy intervention provided by student occupational therapists for 30 minutes a day for eight weeks result in improved resident health status as measured using the EuroQoL-5D Health Questionnaire?

DESCRIPTION OF THE POPULATION TO BE STUDIED, INCLUSION AND STUDY POPULATION

The study population will be residents living at one of the long-term care homes in the Hamilton, St. Joseph's Villa in Dundas, Ontario. These residents will be selected from two home areas with a similar staff complement and similar resident profile. The level of registered and non-registered staff are similar on both units, as are the life enrichment programs offered. Each home area has between 26 and 32 residents. A total of 16 residents will be selected (eight from each home area).

SUBJECT RECRUITMENT

The Resident Assessment Instrument (RAI) Coordinator will identify residents who meet the eligibility criteria and provide the contact details to the primary investigator. The PI will send a letter to potential participants and, when consent is provided, to the families of those residents, describing the study and informing that the PI will be in contact. If, upon contact, the resident agrees, the PI or a co-investigator will meet with the potential participant to inform about the study and request consent. Family members will also be encouraged to also attend.

SAMPLE SIZE

A feasibility sample size will be determined based on the number of residents on each unit who meet the eligibility and inclusion criteria for this study. Based on the 2019-2020 Profile of Residents Ontario in Residential and Hospital-Based Continuing Care 38% of residents scored a 3 or below on the ADL Hierarchy Scale and 66.4% scored a 3 or below on the CPS. Therefore, given the total of residents on both homes areas is 58 a sample size of 16 residents will be chosen. We anticipate, based on this historical Ontario resident data, approximately 22 out of the 58 residents will have an ADL Hierarchy Scale of less or equal to three and 39 residents out of 58 will have a CPS score of less or equal to three.

3.0 STUDY DESIGN The pilot study will be a two-group randomized controlled clinical trial. A total of 16 residents will be allocated in equal proportions to either intervention or no intervention (usual care). Evaluations will be conducted pre-intervention, post-intervention, and at five months post-randomization.

3.1 DESCRIPTION OF METHODOLOGY Investigators will review the Resident Assessment Instrument-Minimum Data Set (RAI-MDS) data provided by the RAI Coordinator at the Long-Term Care Home to identify eligible candidates for occupational therapy intervention based on ADL Long Form, ADL Hierarchy Score and Cognitive Performance Scale. Sixteen residents will be selected (eight from each home area).

A letter and information flyer about the study will be sent to residents and family members (as appropriate) explaining this protocol to those residents eligible to participate. The primary investigator (DCE) and student investigators will obtain verbal and written consent from residents or their designate to participate.

Baseline data will be collected using the following measures:

* Modified Barthel Index
* EuroQoL-5D Health Questionnaire

3.2 RANDOMIZATION

Residents who meet study eligibility criteria and provide consent to participate will be randomly assigned to either the control or intervention group with a 1:1 allocation as per a computer-generated randomisation schedule stratified by baseline score ADL Hierarchy and ADL Long Form Score completed within 5 months of the intervention planned timeframe.

3.3 BLINDING

Once residents are randomly allocated, the Modified Barthel Index and EQ-5D-5L will be administered to all residents by two independent assessors at week one and again at week eight. The assessors will be blinded to the resident's allocation group. Student investigators will not have access to the baseline data. They will only be provided the names of the resident who have been randomized to the intervention group to receive occupational therapy services.

3.4 INTERVENTION The student investigators will complete an initial OT assessment based on a thorough chart review and observation of the participants self-care routine (bathing, dressing, grooming, toileting, eating and mobility) during week one of their eight-week placement clinical placement. Next, the student OTs will conduct an initial assessment using the Canadian Model of Occupational Performance Measure (COPM). Then, based on goals identified by the resident, the student occupational therapists will share their findings based on their chart review, observation of resident performance, and information gathered during the initial assessment with members of the care team.

Next, in collaboration with the resident and the team, the student OT will establish resident-centered goals and develop a targeted intervention plan to address performance issues identified by residents in areas of daily living. The resident will receive approximately 30 minutes a day of direct student OT service delivery. Additional intervention may be delivered through an indirect, collaborative, or consultative service delivery model. Students will use a workload measurement tool to track the amount of time and types of intervention provided to these residents. The intervention will be delivered by two pairs student occupational therapy students under the direction of a registered OT. Student OTs will have access to Point Click Care and will document daily and will be required to document indirect and non-direct time for each resident.

3.5 USUAL CARE

Those residents allocated to the control group will continue to receive usual care. Usual care is defined as an average of four hours of direct care from nurses and personal support workers. Direct care hands-on care that includes personal care, such as feeding, bathing, dressing, and other medical/therapeutic tasks (Ontario Ministry of Long-Term Care, 2020). All residents will continue to have access to 24-hour nursing and personal care in addition to access to all usual programming, including recreation and physiotherapy services.

ELIGIBILITY:
Inclusion Criteria:

Residents eligible for the trial must comply with all the following at randomization:

1. Current admission to St. Joseph's Villa as a long-term care resident.
2. An Activities of Daily Living (ADL) Self-Performance Hierarchy Scale of 4 out of 6 or lower. Higher scores indicate greater decline (progressive loss) in ADL performance.
3. ADL Long Form score of 22 out of 28 or lower. Higher scores indicate more dependence in ADL.
4. Cognitive Performance Scale (CPS) score between 0-3 out of 6 within the last three months. Higher scores indicate more severe cognitive impairment.
5. Individuals can respond or have a caregiver who is able to respond to the EuroQoL-5D Health Questionnaire.
6. Individuals or their proxy are willing to provide consent to participate.

Exclusion Criteria:

1. Residents with a Change in Health, End-Stage Disease and Signs and Symptoms (CHESS) score of equal to 4 or greater on their last assessment, completed within the last three months. This assessment completed for all residents by nursing staff every three months. Higher scores indicate higher levels of medical complexity and are associated with adverse outcomes

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
Modified Bathel Index (MBI) | eight weeks (between July 1st and August 26th, 2022)
  The MBI is a measure of activities of daily living, which shows the degree of independence of a patient from any assistance. It covers 10 domains of functioning (activities): bowel control, bladder control, as well as help with grooming, toilet use, feeding, transfers, walking, dressing, climbing stairs, and bathing. The scoring for the MBI is out of 100. A higher score indicates a greater degree of independence.

SECONDARY OUTCOMES:
EuroQoL-5D | Eight weeks between July 1st and August 26th, 2022
  The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health. The EQ-5D questionnaire also includes a Visual Analog Scale (VAS), by which respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Perrett, Principal Investigator — McMaster University
Locations (1):
- McMaster University, School of Rehabilitation Science, Dundas, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
The plan is to publish the pilot protocol and findings of the pilot student.
Supporting Information: Study Protocol
Time Frame: The data will become available in August, 2022